CLINICAL TRIAL: NCT05291104
Title: Dietary Allowance of Methyl Donor Nutrients to Minimize Risks of Non-alcoholic Fatty Liver Progression: Novel Diagnostic and Therapeutic Markers in Metabolomics of Gut Microbiome/Host Methyl Nutrition and the Working Mechanisms
Brief Title: Dietary Allowance of Methyl Donor Nutrients to Minimize Risks of Non-alcoholic Fatty Liver Progression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fu Jen Catholic University Hospital (Other)
Responsible Party: Principal Investigator, Rwei-Fen Syu Huang, Professor, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C108076
Record Dates: First submitted 2022-03-10; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Methyl nutrients; Non-alcoholic fatty liver; Gut-liver axis; Metabolomics
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Folic Acid; Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (No Intervention): Interventions are not received any treatments.
- Intervention (Experimental): Interventions are received folic acid or choline
  Interventions: Dietary Supplement: Folic acid, choline chloride

INTERVENTIONS:
Dietary Supplement: Folic acid, choline chloride — In this study, we divide intervention group into two groups which received folic acid (FA) or choline chloride (CC) supplement. Each subgroups contain 20 subjects, including 10 men and women. According to Recommended Daily Nutrient Allowance, FA recommended intake is 400 ug / day and choline recommended intake in men and women is 450 and 390 mg / day. From phase 1 to phase 3 stage, for every 10 days, subjects are given 2-fold, 4-fold and 8-fold recommended intake dose of FA or CC. All supplement solve in 240 ml cranberry juice.
  Arms: Intervention

SUMMARY:
Investigate the methyl donors requirement of NAFLD patients to correct the malnutrition, lipid-toxicity, microbiota dysfunction, and metabolomics biomarkers.

DETAILED DESCRIPTION:
Folate/choline/betaine, service as a methyl-donor nutrients, are essential nutrients involving in hepatic one-carbon and bioenergetic metabolism. Methyl-donor nutrients deficiency cause liver and muscle dysfunction as result of non-alcoholic fatty liver diseases (NAFLD) and its progressive lesions of steatohepatitis (NASH), fibrinogen cirrhosis and hepatoma. As methyl-donor nutrients intakes in Taiwanese population are highly insufficient, the dietary requirement of methyl-donor nutrients upon genetic, epigenetic and microbiota interaction to prevent or/and co-therapy of NAFLD progression is currently not known. In this study, we investigate whether intervention of methyl-donor nutrients improve or retard NAFLD progress. NAFLD patients are randomly divided into three groups and received placebo, folic acid, or choline, respectively. From first day to ten day, interventions are given double recommended daily intake dose of folic acid or double adequate Intakes dose of choline, then continuing with four times, and eight times dose for every 10 days. All supplements solve in cranberry juice. At the end of every ten days intervention prior, interventions are measurement of weight and body fat, and collection of blood and feces. The primary outcome measures are described to decreased body weight or body fat, improvement of liver function and fatty liver, and increasing methyl-donor nutrients levels.

ELIGIBILITY:
Inclusion Criteria:

* NAFLD/NASH patients
* Folate levels in plasma < 6 ng/mL or choline levels in plasma < 5 micromol per liter
* Folate intake < estimated average requirement or choline intake < 50% adequate Intakes
* Homocysteine levels in plasma > 9 micromol per liter

Exclusion Criteria:

* Asymptomatic carrier of hepatitis B and C
* Liver disease except NAFLD
* Taking drugs that causes fatty liver
* Inflammation about stomach or intestines
* Pregnancy
* Cancer except liver cancer
* Heart disease, vascular disease, or psychosis
* Intake alcohol over 100 g or unaccessible intake alcohol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Liver fat proportion | One month
  To estimate hepatic fat content, interventions are detected fat content in liver by using MRI or abdominal ultrasound. We assume changing liver fat proportion after finishing intervention.
Improvement liver dysfunction progress | One month
  To estimate liver dysfunction, we detect biochemical markers in plasma, including alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, and glutamyl transpeptidase. After finishing intervention, we assume improving liver function.
Body fat percentage | One month
  Body fat percentage are measured by using electronic body fat meter. Body fat percentage change after intervention.
Plasma methyl nutrients levels | One month
  Folate and choline concentration in plasma are detected to refer methyl nutrients levels. Methyl nutrients levels change after finishing intervention.

SECONDARY OUTCOMES:
Change microbiota | One month
  After intervention change microbiota to improve NAFLD

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Shun Lin, Ph.D, Principal Investigator — Fu Jen Catholic University
Locations (1):
- Taipei Hospital, Ministry of Health and Welfare, New Taipei City, Taiwan